CLINICAL TRIAL: NCT01505777
Title: Exploratory Clinical Study to Evaluate the Optimal Dosage of Mosapride and Probiotics in Irritable Bowel Syndrome Without Predominant Diarrhea: Double Blinded, Randomized, Placebo Drug Controlled, Parallel Designed, Multi-centered, Phase 2 Study
Brief Title: Exploratory Clinical Study to Evaluate the Optimal Dosage of Mosapride and Probiotics in Irritable Bowel Syndrome Without Predominant Diarrhea
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HM-MEMO-201
Record Dates: First submitted 2012-01-03; First posted 2012-01-09 (Estimated); Last update posted 2013-04-05 (Estimated); Status verified 2013-04

CONDITIONS: Irritable Bowel Syndrome Without Diarrhea
Keywords: irritable bowel syndrome without predominant diarrhea; Probiotics(Medirac) 10/mosapride 10mg; Probiotics(Medirac) 15/mosapride 10mg; Probiotics(Medirac) 15/mosapride 15mg; Probiotics(Medirac) 30/mosapride 15mg; Probiotics(Medirac) placebo/mosapride placebo
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Probiotics(Medirac) 10/mosapride 10mg (Experimental)
  Interventions: Drug: Probiotics (Medirac)
- Probiotics(Medirac) 15/mosapride 10mg (Experimental)
  Interventions: Drug: Probiotics (Medirac)
- Probiotics(Medirac) 15/mosapride 15mg (Experimental)
  Interventions: Drug: Probiotics (Medirac)
- Probiotics(Medirac) 30/mosapride 15mg (Experimental)
  Interventions: Drug: Probiotics (Medirac)
- Probiotics(Medirac) placebo/mosapride placebo (Placebo Comparator)
  Interventions: Drug: Probiotics (Medirac) placebo/mosapride placebo

INTERVENTIONS:
Drug: Probiotics (Medirac) — 10/mosapride 10mg three times a day, P.O. 4week
  Arms: Probiotics(Medirac) 10/mosapride 10mg
Drug: Probiotics (Medirac) — 15/mosapride 10mg three times a day, P.O. 4week
  Arms: Probiotics(Medirac) 15/mosapride 10mg
Drug: Probiotics (Medirac) — 15/mosapride 15mg three times a day, P.O. 4week
  Arms: Probiotics(Medirac) 15/mosapride 15mg
Drug: Probiotics (Medirac) — 30/mosapride 15mg three times a day, P.O. 4week
  Arms: Probiotics(Medirac) 30/mosapride 15mg
Drug: Probiotics (Medirac) placebo/mosapride placebo — three times a day, P.O. 4week
  Arms: Probiotics(Medirac) placebo/mosapride placebo

SUMMARY:
The purpose of this study is to Evaluate the Optimal Dosage of Mosapride (Medirac) and Probitics in Irritable Bowel Syndrome Without Predominant Diarrhea.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-75 years who satisfied RomeIII criteria for the diagnosis of IBS
* Signed informed consent

Exclusion Criteria:

* IBS-D
* evidence of cathartic colon or history laxative abuse

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2011-05; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in patient's overall satisfaction relief over 4 weeks of treatment of IBS symptoms | baseline and 4 week

SECONDARY OUTCOMES:
Change from Baseline in improvment of abdominal discomfort, pain, bloating, stool frequency, stool consistency, straining urgency over 4 weeks of treatment and during each week(4 weeks,6 weeks) | baseline and 4 weeks, 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hyo Jin Park, M.D., Ph.D., Principal Investigator — Gangnam Severance Hospital
Locations (1):
- 16 institutions including Gangnam Severance hospital, Seoul, South Korea

REFERENCES:
- [Derived] Choi CH, Kwon JG, Kim SK, Myung SJ, Park KS, Sohn CI, Rhee PL, Lee KJ, Lee OY, Jung HK, Jee SR, Jeen YT, Choi MG, Choi SC, Huh KC, Park H. Efficacy of combination therapy with probiotics and mosapride in patients with IBS without diarrhea: a randomized, double-blind, placebo-controlled, multicenter, phase II trial. Neurogastroenterol Motil. 2015 May;27(5):705-16. doi: 10.1111/nmo.12544. Epub 2015 Mar 25. PMID 25809913